CLINICAL TRIAL: NCT05402735
Title: Value of Uric Acid as Early Predictor of Lupus Nephritis in Assiut University Hospital
Brief Title: Value of Uric Acid as Early Predictor of Lupus Nephritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman gamal neyaz, principle investigator, Assiut University
Other Study IDs: Serum uric acid in SLE
Record Dates: First submitted 2022-05-29; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Uric Acid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Serum uric acid level — Serum uric acid level

SUMMARY:
The aim of the present work is to determine the role of uric acid as a predictor and prognostic factor in the development of lupus nephritis.

DETAILED DESCRIPTION:
Systemic Lupus Erythematosus (SLE) is a systemic autoimmune disorder identified by the production of autoantibodies and immune complex deposition [1]. It presents with a variety of unpredictable flares of disease activity and irreversible organ damage [2]. Half or more (45%-85%) of patients with SLE will develop Lupus Nephritis (LN) over the course of their lifetime, which is a major concern [3,4]. Despite advanced immunosuppressive therapy, the 5-year survival rate of SLE patients with severe renal damage (11%-33%) is usually very low [5].

Hence, early prediction and diagnosis of LN are of great value. So far, renal biopsy remains to be the gold standard tool for diagnosis of LN [6] and assumes a vital role in its management and prognosis. However, renal biopsy can have various complications including hemorrhage and infection. Besides, some patients have contraindications for renal biopsy, which indicates the requirement for noninvasive markers for evaluating renal dysfunction and its grade [7].

- Elimination of serum uric acid (SUA), the circulating endproduct of purine metabolism, occurs via both renal and extrarenal (gastrointestinal tract) pathways [8]. Kang and colleagues [9] have reported that elevated serum uric acid may also be a risk factor for progression of renal disease, in spite of the fact that it is considered as one of the markers of renal dysfunction. Elevated serum uric acid itself can lead to kidney damage without the deposition of uric acid crystals as reported in different studies [10]. Other studies strongly suggest to consider the concept of asymptomaticity for chronic hyperuricemia and hence to check the normal level of serum uric acid levels [11].

Hyperuricemia can be observed in patients with diabetic nephropathy , IgA nephropathy , metabolic syndrome and cardiovascular diseases [12,13,14,15]. In addition, a noteworthy positive relationship was detected between serum level of uric acid and new onset lupus nephritis. Elevated sUA has been observed as an independent risk factor for the development of LN . The correlation between sUA and the degree of renal dysfunction in LN patients was previously analyzed but in a few studies as in Calich and colleagues study who reported an association between lupus nephritis and high serum UA . Therefore the aim of the current study was to evaluate serum uric acid level and detect if hyperuricemia can independently predict and affect prognosis of LN among SLE patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients fulfilled the European League Against Rheumatism (EULAR) and the American college of rheumatology (ACR)

Exclusion Criteria:

* Exclusion criteria were the use of diuretics, aspirin, cyclosporine, or any drugs affect level of uric acid Also exlude patients with hypertension, diabetes , dyslipidemia and obesity

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients fulfilled the European League Against Rheumatism (EULAR) and the American college of rheumatology (ACR)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2023-07-12 (Estimated); Study Completion 2023-08-25 (Estimated)

PRIMARY OUTCOMES:
Value of uric acid as early predictor of lupus nephritis in Assiut University hospital | 1 year
  The aim of the present work is to determine the role of uric acid as a predictor and prognostic factor in the development of lupus nephritis.
  The aim of the present work is to determine the role of uric acid as a predictor and prognostic factor in the development of lupus nephritis.

CONTACTS AND LOCATIONS:
Locations (1):
- assuit University, Asyut, Egypt

REFERENCES:
- [Background] Yuan W, DiMartino SJ, Redecha PB, Ivashkiv LB, Salmon JE. Systemic lupus erythematosus monocytes are less responsive to interleukin-10 in the presence of immune complexes. Arthritis Rheum. 2011 Jan;63(1):212-8. doi: 10.1002/art.30083. PMID 20954190
- [Background] Borchers AT, Leibushor N, Naguwa SM, Cheema GS, Shoenfeld Y, Gershwin ME. Lupus nephritis: a critical review. Autoimmun Rev. 2012 Dec;12(2):174-94. doi: 10.1016/j.autrev.2012.08.018. Epub 2012 Sep 8. PMID 22982174
- [Background] Zubair A, Frieri M. Lupus nephritis: review of the literature. Curr Allergy Asthma Rep. 2013 Dec;13(6):580-6. doi: 10.1007/s11882-013-0394-4. PMID 24234325
- [Background] Koutsokeras T, Healy T. Systemic lupus erythematosus and lupus nephritis. Nat Rev Drug Discov. 2014 Mar;13(3):173-4. doi: 10.1038/nrd4227. Epub 2014 Feb 14. No abstract available. PMID 24525782
- [Background] Cameron JS, Hicks J. The introduction of renal biopsy into nephrology from 1901 to 1961: a paradigm of the forming of nephrology by technology. Am J Nephrol. 1997;17(3-4):347-58. doi: 10.1159/000169122. PMID 9189255
- [Background] Xie T, Chen M, Tang X, Yin H, Wang X, Li G, Li J, Zuo X, Zhang W. Hyperuricemia is an independent risk factor for renal pathological damage and poor prognosis in lupus nephritis patients. Zhong Nan Da Xue Xue Bao Yi Xue Ban. 2016 Oct 28;41(10):1052-1057. doi: 10.11817/j.issn.1672-7347.2016.10.007. PMID 27807327
- [Background] Kang DH, Nakagawa T, Feng L, Watanabe S, Han L, Mazzali M, Truong L, Harris R, Johnson RJ. A role for uric acid in the progression of renal disease. J Am Soc Nephrol. 2002 Dec;13(12):2888-97. doi: 10.1097/01.asn.0000034910.58454.fd. PMID 12444207
- [Background] Desideri G, Castaldo G, Lombardi A, Mussap M, Testa A, Pontremoli R, Punzi L, Borghi C. Is it time to revise the normal range of serum uric acid levels? Eur Rev Med Pharmacol Sci. 2014;18(9):1295-306. PMID 24867507
- [Background] Mazzali M, Hughes J, Kim YG, Jefferson JA, Kang DH, Gordon KL, Lan HY, Kivlighn S, Johnson RJ. Elevated uric acid increases blood pressure in the rat by a novel crystal-independent mechanism. Hypertension. 2001 Nov;38(5):1101-6. doi: 10.1161/hy1101.092839. PMID 11711505
- [Background] Liu P, Chen Y, Wang B, Zhang F, Wang D, Wang Y. Allopurinol treatment improves renal function in patients with type 2 diabetes and asymptomatic hyperuricemia: 3-year randomized parallel-controlled study. Clin Endocrinol (Oxf). 2015 Oct;83(4):475-82. doi: 10.1111/cen.12673. Epub 2014 Dec 29. PMID 25400252
- [Background] Cheng GY, Liu DW, Zhang N, Tang L, Zhao ZZ, Liu ZS. Clinical and prognostic implications of serum uric acid levels on IgA nephropathy: a cohort study of 348 cases with a mean 5-year follow-up. Clin Nephrol. 2013 Jul;80(1):40-6. doi: 10.5414/CN107813. PMID 23391320
- [Background] Li C, Hsieh MC, Chang SJ. Metabolic syndrome, diabetes, and hyperuricemia. Curr Opin Rheumatol. 2013 Mar;25(2):210-6. doi: 10.1097/BOR.0b013e32835d951e. PMID 23370374
- [Background] Sertoglu E. Serum uric acid: an independent predictive marker for coronary artery disease. Clin Rheumatol. 2015 Sep;34(9):1659. doi: 10.1007/s10067-015-2919-9. Epub 2015 Mar 22. No abstract available. PMID 25796387